CLINICAL TRIAL: NCT02025907
Title: A Randomized, Double-blind, Placebo Controlled, 2-arm, Parallel-group, 26-week, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin in the Treatment of Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin and Sitagliptin Therapy
Brief Title: A Study to Evaluate the Efficacy and Safety of the Addition of Canagliflozin in Participants With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin and Sitagliptin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR103477; 2013-004819-40 (EudraCT Number); 28431754DIA4004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Results first posted 2016-09-02 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Canagliflozin; Hemoglobin A1c; Metformin; Sitagliptin; T2DM; JNJ-28431754
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canagliflozin (JNJ-28431754) (Experimental): Each participant will receive canagliflozin (JNJ-28431754) 100 mg once daily during the first 6 weeks, then the dose may be increased to 300 mg once daily.
  Interventions: Drug: Canagliflozin, 100 mg; Drug: Canagliflozin, 300 mg
- Placebo (Placebo Comparator): Each participant will receive placebo (inactive medication) once daily for 28 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin, 100 mg — One 100 mg capsule taken orally (by mouth) once daily.
  Arms: Canagliflozin (JNJ-28431754)
Drug: Canagliflozin, 300 mg — One 300 mg capsule taken orally (by mouth) once daily.
  Arms: Canagliflozin (JNJ-28431754)
Drug: Placebo — One placebo capsule taken orally (by mouth) once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of canagliflozin (JNJ-28431754) compared to placebo in the treatment of participants with Type 2 Diabetes Mellitus (T2DM), who have inadequate glycemic control on maximally or near-maximally effective doses of metformin and sitagliptin.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), placebo-controlled (an inactive substance that is compared with a study drug, to test whether the study drug has a real effect), multicenter study of efficacy, safety, and tolerability of canagliflozin in participants with T2DM, who have inadequate glycemic (blood sugar) control on maximally or near-maximally effective doses of metformin >=1500 mg/day and sitagliptin 100 mg/day. Approximately 200 participants will be randomly assigned to 1 of 2 treatment groups in 1:1 ratio for 26 weeks. During the study the participants will be also provided with diet and exercise counseling (standardized non-pharmacological therapy).

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of type 2 diabetes mellitus
* Must have a screening HbA1c of >=7.5% to <=10.5%
* Must be on metformin >=1500 mg/day and sitagliptin 100 mg/day (or equivalent fixed dose combination) at a stable dose for at least 12 weeks before screening

Exclusion Criteria:

* History of diabetic ketoacidosis or T1DM, hereditary glucose-galactose malabsorption or primary renal glycosuria
* A myocardial infarction, unstable angina, revascularization procedure or cerebrovascular accident within 12 weeks before screening
* eGFR <60 ml/min/1.73m2, or serum creatinine >=1.4 mg/dL for men and >=1.3 mg/dL for women
* Known significant liver disease (eg, acute hepatitis, chronic active hepatitis, cirrhosis)
* Major surgery (ie, requiring general anesthesia) within 12 weeks before screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (57):
- United States (30):
  - Montgomery, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Northridge, California
  - Norwalk, California
  - Rancho Cucamonga, California
  - San Ramon, California
  - Aurora, Colorado
  - Denver, Colorado
  - Littleton, Colorado
  - Cooper City, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Atlanta, Georgia
  - Perry, Georgia
  - Shawnee Mission, Kansas
  - Marrero, Louisiana
  - Metairie, Louisiana
  - Metarie, Louisiana
  - Rockville, Maryland
  - Jackson, Mississippi
  - Picayune, Mississippi
  - St Louis, Missouri
  - Nashua, New Hampshire
  - Albuquerque, New Mexico
  - Albany, New York
  - Arlington, Texas
  - San Antonio, Texas
  - Sugarland, Texas
  - Bountiful, Utah
- Australia (10):
  - Coffs Harbour
  - Freemantle
  - Geelong
  - Heidelberg
  - Herston
  - Melbourne
  - Merewether
  - Sherwood
  - Sydney
  - Wollongong
- Canada (3):
  - Brampton, Ontario
  - Hawkesbury, Ontario
  - Toronto, Ontario
- France (7):
  - La Rochelle Cedex 1 Poitou-Cha
  - La Tronche
  - Nancy
  - Narbonne
  - Nice
  - Paris
  - Vénissieux
- Germany (7):
  - Freiburg im Breisgau
  - Fulda
  - Hamburg
  - Münster
  - Neuwied
  - Pirna
  - Speyer

REFERENCES:
- [Derived] Cai J, Delahanty LM, Akapame S, Slee A, Traina S. Impact of Canagliflozin Treatment on Health-Related Quality of Life among People with Type 2 Diabetes Mellitus: A Pooled Analysis of Patient-Reported Outcomes from Randomized Controlled Trials. Patient. 2018 Jun;11(3):341-352. doi: 10.1007/s40271-017-0290-4. PMID 29313267

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was randomized at 2 different sites (once to placebo and once to canagliflozin) and was therefore counted twice in the total number of randomized participants. The participant was withdrawn from the study and not included in any efficacy or safety analyses.
Groups:
- Placebo: Participants administered with placebo (inactive medication) once daily for 26 weeks.
- Canagliflozin: Participants administered canagliflozin (JNJ-28431754) 100 milligram (mg) titratable to 300 mg once daily for 26 weeks.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin
Started | 108 (Participant flow is presented for safety population.) | 108 (Participant flow is presented for safety population.)
Completed | 81 | 96
Not Completed | 27 | 12
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 15 | 8
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Potential misconduct,GCPcompliance issue | 2 | 1

BASELINE CHARACTERISTICS:
Population: mITT (modified intent-to-treat) population included all randomized participants who received at least 1 dose of double-blind study drug. A total of 3 participants were excluded from the mITT population due to potential misconduct and GCP compliance issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin | Total
Number analyzed (Participants) | 106 | 107 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.14) | 57.4 (9.28) | 57.4 (9.69)
Gender [Count of Participants; unit: Participants]
  Female | 51 | 41 | 92
  Male | 55 | 66 | 121
Region of Enrollment [Number; unit: participants]
  Australia | 13 | 22 | 35
  Canada | 16 | 23 | 39
  France | 10 | 6 | 16
  Germany | 16 | 13 | 29
  United States | 51 | 43 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26
Time Frame: Baseline and Week 26
Population: mITT population included all randomized participants who received at least 1 dose of double-blind study drug. A total of 3 participants were excluded from the mITT population due to potential misconduct and GCP compliance issues. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo | Canagliflozin
Number analyzed (Participants) | 94 | 99
percentage of glycosylated hemoglobin | -0.01 (0.119) | -0.91 (0.113)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter
Arm/Group | Placebo | Canagliflozin
Number analyzed (Participants) | 104 | 103
millimoles per liter | -0.14 (0.281) | -1.65 (0.264)

3. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 26
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Canagliflozin
Number analyzed (Participants) | 104 | 103
percent change | -1.60 (0.337) | -3.35 (0.324)

4. Secondary Outcome: Percentage of Participants With HbA1c Less Than (<) 7.0 Percent at Week 26
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Canagliflozin
Number analyzed (Participants) | 82 | 96
percentage of participants | 12.2 | 32.3

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 26
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin
Number analyzed (Participants) | 104 | 103
millimeter of mercury (mmHg) | 0.09 (1.123) | -5.76 (1.078)

ADVERSE EVENTS:
Time Frame: From Baseline, up to end of treatment (Approximately 31 weeks)
Description: Safety population included all randomized participants who received at least 1 dose of double-blind study drug and 3 participants who were excluded from the mITT population due to potential misconduct and GCP compliance issues.
Arm/Group | Placebo | Canagliflozin
Serious Adverse Events (participants affected / at risk) | 2/108 | 2/108
Other Adverse Events (participants affected / at risk) | 16/108 | 18/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Canagliflozin (N=108)
Angina Unstable (Cardiac disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Canagliflozin (N=108)
Nasopharyngitis (Infections and infestations) | 6 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Depression (Psychiatric disorders) | 0 | 3
Polyuria (Renal and urinary disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.